CLINICAL TRIAL: NCT00001454
Title: Endometrial Mediators of Gonadal Steroid Action
Brief Title: Hormonal Effects on the Uterus and Endometrium
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 950110; 95-CH-0110
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2019-12-16 (Actual); Status verified 2015-07-27

CONDITIONS: Pregnancy
Keywords: Estrogen; Progesterone; Menses; Endometrium; Normal Volunteer

SUMMARY:
Endometrium is the lining of the uterus. It is where the fertilized egg normally implants during pregnancy.

This study was designed to better understand the way(s) that female sex hormones (estrogen and progesterone) cause the uterus to grow and develop. It is known that these hormones are necessary to prepare the uterus for pregnancy, but the way the hormones work is unknown.

Researchers would like to identify the genes that are affected by female sex hormones by using a variety of tests (in situ hybridization, immunohistochemistry, and culture of human endometrium).

Researchers will select women who have regular monthly menstrual cycles and study them for two cycles;

1. <TAB>The first cycle (PRE-BIOPSY CYCLE) will include daily measurements of the patient's body temperature and progesterone measurements during the last 14 days (luteal phase) of the menstrual cycle.
2. <TAB> The second cycle (BIOPSY CYCLE) will include measurements of urinary luteinizing hormone (LH) to determine the day of the LH surge. Luteinizing hormone is the hormone that causes the ovary to release the developed egg. Ovarian ultrasounds will be performed before the biopsy to determine development of the egg. Blood tests will be taken on the day of the biopsy to have an overall idea of the hormones circulating in the patient's blood. An endometrial biopsy will be taken at one of three possible times to identify endometrial products under conditions of estrogen, estrogen/progesterone, or steroid hormone withdrawal.<TAB>

DETAILED DESCRIPTION:
Estrogen and progesterone induce characteristic and predictable morphological changes in the endometrium that are required for successful implantation and pregnancy. The mechanism(s) by which estrogen and progesterone exert these effects on the endometrium is not known. This is a tissue collection protocol to obtain endometrium and/or menstrual effluent from normally cycling women, women with endometriosis and women with infertility.

This tissue will be used for future studies intended to understand gonadal steroid action on the endometrium We propose to identify peptides that are induced by endogenous estrogen and progesterone using in situ hybridization, immunohistochemistry, microarray analysis and/or culture of human endometrium obtained at hormonally different times of the cycle. Regularly cycling women not at risk for pregnancy will be studied for two menstrual cycles. The first, pre-biopsy cycle, will be characterized by daily basal body temperature measurements and a luteal phase progesterone measurement. During the biopsy cycle, urinary LH measurements will be performed to determine the day of the LH surge. Ovarian ultrasounds to assess follicular development will be performed before biopsy. Blood will be obtained on the day of the biopsy to characterize the hormonal mileau. An endometrial biopsy will be obtained either in the early follicular phase (at a follicular diameter of less than 8 mm), the late follicular phase (follicular diameter greater than 14 mm) or in the mid-(luteal phase day 6-8) or late (luteal phase day 12 - 14) luteal phase, to allow identification of endometrial products under conditions of estrogen, estrogen/progesterone and steroid withdrawal. Alternatively, endometrial tissue may be obtained from normal women and those with endometriosis at the time of menses using a cup-shaped intravaginal collecting device. Additionally, women with infertility possibly related to endometrial dysfunction will be studied in the luteal phase.

ELIGIBILITY:
* INCLUSION CRITERIA:

Healthy volunteers will be in excellent health.

Only women with regular menstrual cycles (every 26-35 days) using mechanical (condoms, diaphragm) or sterilization methods of contraception will be included.

Only women with a negative pregnancy test, normal physical examination and laboratory results, and a luteal phase progesterone value of greater than 4 ng/mL will be entered into this study.

Women with endometriosis will be recruited from those with histologically-proven endometriosis. Except for this diagnosis they will meet criteria for healthy volunteers as stated above.

Women may participate in the study on more than one occasion, but biopsies may not be performed in a "baseline" cycle.

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 129 (Actual)
Dates: Start 1995-04-21; Study Completion 2015-07-27

CONTACTS AND LOCATIONS:
Overall Officials: Lynnette K Nieman, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Sokolov BP, Prockop DJ. A rapid and simple PCR-based method for isolation of cDNAs from differentially expressed genes. Nucleic Acids Res. 1994 Sep 25;22(19):4009-15. doi: 10.1093/nar/22.19.4009. PMID 7524031
- [Background] Jones GS. The clinical evaluation of ovulation and the luteal phase. J Reprod Med. 1977 Mar;18(3):139-42. No abstract available. PMID 853495
- [Background] Batista MC, Cartledge TP, Merino MJ, Axiotis C, Platia MP, Merriam GR, Loriaux DL, Nieman LK. Midluteal phase endometrial biopsy does not accurately predict luteal function. Fertil Steril. 1993 Feb;59(2):294-300. PMID 8425621